CLINICAL TRIAL: NCT00004241
Title: A Phase I Trial of Weekly 17-Allylamino-17 Demethoxygeldanamycin
Brief Title: 17-N-Allylamino-17-Demethoxygeldanamycin in Treating Patients With Advanced Epithelial Cancer, Malignant Lymphoma, or Sarcoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02315; PCI-99-020; U01CA099168 (NIH); CDR0000067486 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-01-28; First posted 2003-01-27 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: AIDS-related Peripheral/Systemic Lymphoma; AIDS-related Primary CNS Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Chondrosarcoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Intraocular Lymphoma; Metastatic Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor; Metastatic Osteosarcoma; Nodal Marginal Zone B-cell Lymphoma; Ovarian Sarcoma; Primary Central Nervous System Non-Hodgkin Lymphoma; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult Soft Tissue Sarcoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Osteosarcoma; Recurrent Small Lymphocytic Lymphoma; Recurrent Uterine Sarcoma; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Mixed Cell Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Adult Hodgkin Lymphoma; Stage IV Adult Immunoblastic Large Cell Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Adult Soft Tissue Sarcoma; Stage IV Adult T-cell Leukemia/Lymphoma; Stage IV Cutaneous T-cell Non-Hodgkin Lymphoma; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Mycosis Fungoides/Sezary Syndrome; Stage IV Small Lymphocytic Lymphoma; Stage IV Uterine Sarcoma; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Chondrosarcoma; Intraocular Lymphoma; Neuroectodermal Tumors, Primitive, Peripheral; Osteosarcoma; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Sarcoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — tanespimycin

ARMS (2):
- Schedule B (tanespimycin) (Experimental): Patients receive 17-AAG IV over 1-2 hours twice weekly for 3 weeks. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: tanespimycin; Other: pharmacological study
- Schedule C (tanespimycin) (Experimental): Patients receive 17-AAG IV over 1-2 hours twice weekly for 2 weeks. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: tanespimycin; Other: pharmacological study

INTERVENTIONS:
Drug: tanespimycin — Given IV
  Other Names: 17-AAG
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
Drugs used in chemotherapy work in different ways to stop cancer cells from dividing so they stop growing or die. This phase I trial is studying the side effects and best dose of 17-N-allylamino-17-demethoxygeldanamycin in treating patients with advanced epithelial cancer, malignant lymphoma, or sarcoma

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the dose-limiting toxicity and maximum tolerated dose of 17-N-allylamino-17-demethoxygeldanamycin (17-AAG) in patients with advanced epithelial cancer, malignant lymphoma, or sarcoma.

II. Determine the significant toxic effects associated with this drug in these patients.

III. Determine the response in patients treated with this drug. IV. Determine the pharmacokinetics of 17-AAG and 17AG in these patients.

OUTLINE: This is a dose-escalation study. Patients receive treatment according to 1 of 2 schedules.

Schedule B: Patients receive 17-N-allylamino-17-demethoxygeldanamycin (17-AAG) IV over 1-2 hours twice weekly for 3 weeks. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Schedule C: Patients receive 17-AAG IV over 1-2 hours twice weekly for 2 weeks. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

In both schedules, cohorts of 3-6 patients receive escalating doses of 17-AAG until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. At least 6 patients receive treatment at the MTD.

PROJECTED ACCRUAL: A maximum of 60 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced epithelial cancer, malignant lymphoma, or sarcoma for which no standard curative therapy exists
* Brain metastases allowed after definitive radiotherapy
* Performance status - ECOG 0-2
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 mg/dL
* SGOT no greater than 2 times normal
* Creatinine no greater than 1.5 mg/dL
* Creatinine clearance at least 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception for at least 1 week before, during, and for at least 2 weeks after study completion
* No active infection
* No other serious concurrent condition
* No prior allergic reaction to egg products
* At least 4 weeks since prior biologic therapy (regional or systemic)
* At least 4 weeks since prior chemotherapy
* See Disease Characteristics
* At least 4 weeks since prior radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 1999-10; Primary Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
MTD defined as the dose level preceding that at which 2 of 6 patients experience dose-limiting toxicity (DLT) assessed using Common Toxicity Criteria version 2.0 | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ramesh Ramanathan, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States